CLINICAL TRIAL: NCT02239263
Title: Investigation of Nucleus 6 Sound Processor Input Processing in Cochlear Implant Recipients.
Brief Title: N6 Input Processing in Traditional CI Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM5555
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Results first posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- N6 Input Processing Features (Experimental)
  Interventions: Device: Nucleus 6 Sound Processor

INTERVENTIONS:
Device: Nucleus 6 Sound Processor

SUMMARY:
The purpose of this study is to evaluate the enhanced signal processing features of the Nucleus 6 Sound Processor on existing Nucleus cochlear implant recipients currently using the Nucleus 5 Sound Processor.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 12 years
* Unilateral cochlear implant recipient (CI24RE, CI500, CI422)
* Minimum of 3 months experience with the N5 sound processor
* Prior documentation of sentence recognition testing in noise at a difficulty of +10 dB SNR or better
* Native English speaker
* Willingness to participate in and comply with all requirements of the protocol

Exclusion Criteria:

* Unrealistic expectations
* Unwillingness to comply with investigational requirements of the protocol
* Additional handicaps that would prevent or restrict participation in the evaluations

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-05; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Rocky Mountain Ear Center, Englewood, Colorado
  - Center for Hearing and Balance, Chesterfield, Missouri
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Houston Ear Research Foundation, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As of the date of database closure, 34 of the 40 enrolled subjects completed Visit Two (endpoint testing).
Groups:
- N6 Input Processing Features - SNR-NR & SCAN: Testing of the Nucleus 6 sound processing Signal to Noise Ratio - Noise Reduction (endpoint 1) and SCAN (endpoint 2)
Period: Overall Study
Arm/Group | N6 Input Processing Features - SNR-NR & SCAN
Started | 40
Completed (6 subjects were programmed with the incorrect settings for testing and therefore were excluded from the final data set.) | 34
Not Completed | 6
Not completed — Protocol Violation | 6

BASELINE CHARACTERISTICS:
Arm/Group | N6 Input Processing Features - SNR-NR & SCAN
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (21.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Endpoint 1: Evaluation of Signal to Noise Ratio - Noise Reduction
Description: Speech understanding in noise using AzBio sentences with and without the SNR - noise reduction algorithm enabled. Speech understanding at a fixed +10 dB signal to noise level in each condition (on/off) is scored as percent correct and then subtracted to demonstrate the percent difference (benefit) in performance of having the algorithm on vs off.
Time Frame: Visit 2, 1 month after baseline testing
Measure: Mean (95% Confidence Interval); unit: difference in percent correct scores
Groups:
- N6 Input Processing Features - SNR: Endpoint 1: Assessment of Nucleus 6 sound processing feature SNR-NR
Arm/Group | N6 Input Processing Features - SNR
Number analyzed (Participants) | 34
difference in percent correct scores | -5.9 [-9.6 to -2.2]

2. Primary Outcome: Endpoint 2: Evaluation of SCAN
Description: Speech understanding in noise using AzBio sentences with and without SCAN algorithm enabled. Speech understanding at a fixed +10 dB signal to noise level in each condition (on/off) is scored as percent correct and then subtracted to demonstrate the percent difference (benefit) in performance of having the algorithm on vs off.
Time Frame: Visit 2, 1 month after baseline testing
Measure: Mean (95% Confidence Interval); unit: difference in percent correct scores
Groups:
- N6 Input Processing Features: Endpoint 1: Assessment of Nucleus 6 sound processing feature SCAN
Arm/Group | N6 Input Processing Features
Number analyzed (Participants) | 34
difference in percent correct scores | -26.9 [-33 to -20.9]

ADVERSE EVENTS:
Groups:
- N6 Input Processing Features - SNR-NR: Testing of the Nucleus 6 sound processing Signal to Noise Ratio - Noise Reduction (endpoint 1)
- N6 Input Processing Features - SCAN: Testing of the Nucleus 6 sound processing SCAN (endpoint 2)
Arm/Group | N6 Input Processing Features - SNR-NR | N6 Input Processing Features - SCAN
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No